CLINICAL TRIAL: NCT04762589
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Assess Efficacy, Long Term Safety and Tolerability of RT001 in Subjects With Amyotrophic Lateral Sclerosis
Brief Title: RT001 in Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biojiva LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RT001-014
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — RT001; Safflower Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo-controlled, double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- RT001 (Experimental): RT001 960 mg capsule. 3 capsules TID for 4 weeks, followed by 3 capsules BID for the remaining 20 weeks.
  Interventions: Drug: RT001
- Placebo (Placebo Comparator): Inactive comparator capsule 960 mg (safflower oil). 3 capsules TID for 4 weeks, followed by 3 capsules BID for the remaining 20 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RT001 — RT001 8.64 g/d (3 capsules TID) for 1 month followed by 5.76 g/d (3 capsules BID) for an additional 5 months
  Other Names: di-deuterated linoleic acid ester
  Arms: RT001
Drug: Placebo — Placebo Comparator: Placebo Inactive comparator capsule 960 mg/capsule: 3 capsules TID for 4 weeks, followed by 3 capsules BID for the remaining 20 weeks.
  Other Names: safflower oil
  Arms: Placebo

SUMMARY:
RT001-014 is a Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Assess Efficacy, Long Term Safety and Tolerability of RT001 in Subjects with Amyotrophic Lateral Sclerosis

DETAILED DESCRIPTION:
Forty subjects at 4 EU sites will undergo baseline examination, and then be randomized 1:1 to receive either RT001 or placebo. Repeat visits will occur every 2 months. The final visit will be at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject with age 20 years to 75 years at the time of signed consent
2. Patients who are defined as "definite ALS," "probable ALS" or "probable-laboratory-supported ALS," met diagnostic criteria revised EL Escorial for Airlie House.
3. ALSFRS-R > 20
4. Patients who can eat a meal, excrete, or move with oneself alone, and do not need assistance in everyday life
5. Patients of less than 3 years after the onset of ALS
6. Subject has an identified, reliable, study partner (e.g., caregiver, family member, social worker, or friend)
7. If patients are duly capable of study consent but are unable to sign by themselves due to aggravation of disease condition, written informed consent can be obtained from a legally authorized representative who can sign on behalf of the patients after confirming the patients' agreement to study participation

Exclusion Criteria:

1. Received treatment with other experimental therapies within the last 30 days prior to the first dose
2. Previously received treatment with RT001
3. Refusal to discontinue fish oils or other oil-based supplements for the duration of the study (Screening till last study procedure completed)
4. SVC < 70 at screening
5. Subject has a feeding tube or the need for a feeding tube is anticipated within the first 24 weeks after enrollment
6. Subject resides at a skilled nursing or dementia care facility, or admission to such a facility is planned during the study period
7. Evidence of any clinically significant neurological disorder other than ALS
8. The subject has a history of or currently has schizophrenia, schizoaffective disorder or bipolar disorder according to DSM-V or ICD-10 criteria
9. The subject has a significant pulmonary disorder not attributed to ALS or who require treatments that might complicate the evaluation of the effect of ALS on respiratory function
10. Subject has had a significant illness or infection requiring medical intervention in the past 30 days
11. Female who is breastfeeding or has a positive pregnancy test
12. Male participant or female participant of childbearing potential, who is sexually active and unwilling/unable to use a medically acceptable and effective double barrier birth control method throughout the study
13. Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to return for visits as scheduled
14. History, within the last 2 years, of alcohol abuse or physical opioid dependence

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the revised ALS Functional Rating Score (ALSFRS-R) at 24 weeks | 24 weeks
  Change from baseline in ALSFRS-R will be compared for the RT001 treated group vs placebo

SECONDARY OUTCOMES:
Composite of Death or a Specified State of Disease Progression | 24 weeks
  Change from baseline in the composite endpoint will be compared for the RT001 treated group vs placebo
Change from Baseline in ALS Assessment Questionnaire (40 Items) (ALSAQ40) | 24 weeks
  Change from baseline in ALSAQ40 will be compared for the RT001 treated group vs placebo
Change from baseline in SVC | 24 weeks
  Change from baseline in SVC will be compared for the RT001 treated group vs placebo
Frequency, severity and relationship to study drug of AEs and SAEs | 24 weeks
  Frequency, severity and relationship to study drug of AEs and SAEs will be compared for the RT001 treated group vs placebo

CONTACTS AND LOCATIONS:
Overall Officials: Leonard van den Berg, MD, Principal Investigator — UMC Utrecht
Locations (4):
- University of Tartu, Tartu, Estonia
- Riga Stradins Universtiy, Riga, Latvia
- UMC Utrecht, Utrecht, Netherlands
- Karolinska, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No